CLINICAL TRIAL: NCT01103791
Title: A Trial to Determine the Maximum Tolerated Dose and Evaluate the Safety and Pharmacokinetics of Docetaxel-PNP, Polymeric Nanoparticle Formulation of Docetaxel, in Subjects With Advanced Solid Malignancies
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Samyang Biopharmaceuticals Corporation (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: DOPNP101
Record Dates: First submitted 2010-04-05; First posted 2010-04-15 (Estimated); Last update posted 2017-05-05 (Actual); Status verified 2017-05

CONDITIONS: Advanced Solid Malignancies

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (6):
- Cohort 1 (Experimental): Docetaxel-PNP 20mg/m2
  Interventions: Drug: Docetaxel-PNP
- Cohort 2 (Experimental): Docetaxel-PNP 35mg/m2
  Interventions: Drug: Docetaxel-PNP
- Cohort 3 (Experimental): Docetaxel-PNP 45mg/m2
  Interventions: Drug: Docetaxel-PNP
- Cohort 4 (Experimental): Docetaxel-PNP 60mg/m2
  Interventions: Drug: Docetaxel-PNP
- Cohort 5 (Experimental): Docetaxel-PNP 75mg/m2
  Interventions: Drug: Docetaxel-PNP
- Cohort 6 (Experimental): Docetaxel-PNP 90mg/m2
  Interventions: Drug: Docetaxel-PNP

INTERVENTIONS:
Drug: Docetaxel-PNP — Docetaxel-PNP, Polymeric Nanoparticle Formulation of Docetaxel

SUMMARY:
This is a phase I trial to determine the maximum tolerated dose and recommended phase II dose of docetaxel-PNP (polymeric nanoparticle formulation of docetaxel) and to evaluate the safety and pharmacokinetics of docetaxel-PNP in subjects with advanced solid malignancies.

ELIGIBILITY:
Inclusion Criteria:

* Patient ages more than 18 years old
* Patient should voluntarily sign a written informed consent before study entry
* Patient historically or cytologically confirmed diagnosis of advanced solid tumor and patient with measurable disease or evaluable disease by RECIST criteria
* Progressive disease with development of new lesions or an increase in preexisting lesions or standard therapy in order to provide clinical benefit does not exist or is no longer effective
* Previous anti-cancer therapies must be completed before 21days of first study dose and Patient must have recovered from any previous therapy
* Patient has an Eastern Cooperative Oncology Group (ECOG) Performance Status 0-1
* Patient has a life expectancy of at least 3 months
* Baseline studies for determining eligibility must be completed within 14 days of first study dose and patient has a adequate organ function including the following:

  * Hb ≥ 10g/dl
  * ANC ≥ 1.5 X 109/L
  * Platelet count ≥ 100 X 109/L
  * Serum total bilirubin ≤ 1.5 mg/dL
  * Serum AST and ALT ≤ 2.5 X UNL
  * Serum ALP ≤ 2.5ⅹUNL
  * Serum creatinine ≤ 1.5 X UNL

Exclusion Criteria:

* Patient has had a major surgery except tumor ablation within 2 weeks before screening visit
* Patient has a brain metastasis with neurologic symptom
* Patient has a sensory neuropathy or motor neuropathy ≥ grade 2 by NCI-CTCAE
* Patient has any serious concurrent disease such as:

Any medical or psychiatric condition that, in the opinion of the investigator, would prohibit the understanding and giving of informed consent Severe cardiovascular disease (e.g. ischemic heart disease requiring medication or myocardial infraction within the past six months, grade 3-4 congestive heart failure defined by the New York Heart Association criteria) Active un controlled infection.

* Patient has hypersensitivity to the Investigational product or their excipients
* Patient has participated in any other clinical trial within 4 weeks before screening visit
* Woman is pregnant or breast feeding
* Subjects who are of childbearing potential who do not use a medically acceptable method of birth control or do not agree to continue use of this method throughout the trial (screening, treatment period, and 3 weeks from the last done). A negative pregnancy test (urine or serum) should be documented within 14 days prior to initiation of trial medication for women of childbearing potential who have not been amenorrheic for at least 12 months prior to registration into the trial or surgically sterile (bilateral tubal ligation, bilateral oophorectomy or hysterectomy). Medically acceptable methods include:

  * Barrier method with spermicide
  * Intrauterine device
  * Complete abstinence, etc.
* Patient who has a history of resistance, intolerance, or no response to Docetaxel therapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 19 (Actual)
Dates: Start 2010-04 (Actual); Primary Completion 2011-09 (Actual); Study Completion 2012-04 (Actual)

PRIMARY OUTCOMES:
The maximum tolerated dose (MTD) of Docetaxel-PNP | up to 6 cycle
  Administration of docetaxel-PNP was well tolerated up 6mg/m² every 3weeks by heavily pretreated patients.
The recommended phase II dose of Docetaxel-PNP | up to 6 cycle
  Futher phase Ⅱ Trials are recommended at this dose level

SECONDARY OUTCOMES:
The Dose Limiting Toxicity (DLT) | up to 6 cycle
The pharmacokinetics of Docetaxel-PNP on Day 1 of 1st cycle (AUC, CL, T1/2, Tmax, Cmax, Vdss) | up to 6 cycle
Objective response rate | up to 6 cycle

CONTACTS AND LOCATIONS:
Overall Officials: Kyung Hae Jung, Ph. D., Principal Investigator — Asan Medical Center
Locations (1):
- Asan Medical Center, Seoul, South Korea